CLINICAL TRIAL: NCT04569929
Title: Clinical Evaluation of Implant Overdentures Fabricated Using 3D -Printing Technology Versus Conventional Fabrication Technique: A Randomized Trial
Brief Title: 3D-printed Implant Overdentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Dina ElAwady, lecturer of Prosthodontics (principal investigator), October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Modern Science and Art Uni
Record Dates: First submitted 2020-09-23; First posted 2020-09-30 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Edentulous Mouth
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): conventionally manufactured Polymethyl Methacrylate (PMMA) mandibular implant overdentures
  Interventions: Other: (DLP)-printed photo-polymerizable PMMA Nextdent mandibular implant overdenture
- intervention (Experimental): digital light processed (DLP)-printed photo-polymerizable PMMA Nextdent mandibular implant overdentures
  Interventions: Other: (DLP)-printed photo-polymerizable PMMA Nextdent mandibular implant overdenture

INTERVENTIONS:
Other: (DLP)-printed photo-polymerizable PMMA Nextdent mandibular implant overdenture — The bite registration records with their corresponding master casts were digitalized using an extra oral desktop 3D scanner (3shape D850) and then stored as standard triangulation language (STL) files (Figure 1). The STL files were then imported to Dental system PREMIUM3 design software (3Shape Dental System 2018) for model analysis, surveying and blocking out, designing full permanent denture bases, and for virtual teeth set-up following the recorded inter-arch space

SUMMARY:
A randomized clinical trial (RCT) was designed. Fourteen completely edentulous participants were randomly allocated into two equal groups. All participants received two implants in the inter-foraminal area with ball attachments. Participants in the control group were rehabilitated with conventionally manufactured Polymethyl Methacrylate (PMMA) maxillary complete denture and mandibular implant overdentures while participants in intervention group received digital light processed (DLP)-printed photo-polymerizable PMMA Nextdent maxillary complete denture and mandibular implant overdentures. Follow-up appointments were scheduled at 3,6, and 12 months where data of Oral Health Impact Profile 19(OHIPEDENT19) was used to assess the OHRQoL (oral health related quality of life). In addition, denture retention was measured using digital force gauge device. Data were collected and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous
* ranging in age from 50 to 65 years
* Angle's class I skeletal relationship, normal facial symmetry.
* Adequate quantity of bone (class IV -VI ) and quality (classes 1 - 3 ) in the mandibular inter-foraminal area to accommodate standard implants of at least 11 mm length and 3.7 mm diameter
* appropriate inter-arch space of at least 15 mm (class I ) to accept all types of tested dentures

Exclusion Criteria:Metabolic disorders affecting osseointegration such as hepatic disorders

* osteoporosis and diabetes mellitus.
* Temporomandibular disorders, anticoagulant therapy or bleeding disorders
* sharp mandibular residual ridge or flabby tissues
* neuromuscular disorders, and class II and III Angle's classification skeletal relationship
* Smokers and patients on chemotherapy or radiotherapy or suffering from psychiatric conditions

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
. OHRQoL (oral health related quality of life) | 12 months
  Oral Health Impact Profile 19 (OHIPEDENT19) was used to assess the OHRQoL (oral health related quality of life). The questionnaire was translated to Arabic and validated (S2).24 The profile consisted of 19 questions each with score 0 to 4 (impaired) on Likert scale; accordingly, for each patient the minimum score was 0 and maximum score was 76.

SECONDARY OUTCOMES:
Overdentures' retention | 12 months
  The retention was measured at baseline (day of delivery), three months thereafter, after six months then after 12m by a digital force gauge device (Extech's Model 475055 Digital Force Gauge FLIR Commercial Systems, Inc.) that measures tension or compression force (pull/push) to values of up to 980 Newton.25 The snap hook of the device engaged a screw fixed to the geometric center of denture bases using self-cure acrylic resin. Then pulling action was applied till the denture separation recording the amount of retention in Newton.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Elawady, PHD, Principal Investigator — MSA
Locations (1):
- Msa Uni, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No